CLINICAL TRIAL: NCT02202343
Title: Effectiveness of School-based Health and Nutrition Education to Improve Health and Dietary Practices of Primary School Children From Jimma Zone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jimma University (Other)
Collaborators: World Bank (Other); Ethiopian Public Health Institute (Other Government)
Responsible Party: Principal Investigator, Alemayehu Argaw, Researcher, Jimma University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SHNP/2013
Record Dates: First submitted 2014-07-26; First posted 2014-07-29 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Behaviour
Keywords: Nutrition; Food; Security; School; Health
MeSH Terms: conditions — Behavior | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- School-based health and nutrition education (Experimental)
  Interventions: Behavioral: school based health and nutrition education

INTERVENTIONS:
Behavioral: school based health and nutrition education

SUMMARY:
School based Health and Nutrition Education (SHNE) is a key component of school health and nutrition programs that can address several health and nutrition issues in Ethiopia.

ELIGIBILITY:
Inclusion Criteria:

* Grade 5 to 8

Exclusion Criteria:

* Mental Problem
* Has no Family

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1000 (Actual)
Dates: Start 2013-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Effectiveness of school based health and nutrition education on on health, diet related behavior and food security | 1 year

SECONDARY OUTCOMES:
impacts of health and nutritional education on food hygiene and reproductive health | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Alemayehu A Alemayehu, Researcher, Principal Investigator — Jimma University
Locations (1):
- Jimma University, Jimma, Oromiya, Ethiopia